CLINICAL TRIAL: NCT01149642
Title: Phase III Multicenter, Randomised and Double-blind Study Comparing an Oral Immunomodulatory Solution Versus a Placebo in Preventing Severe Acute Mucositis in Head and Neck Cancer Patients Treated Surgically and Concomitantly With Radiochemotherapy
Brief Title: Randomised Study of Mucositis Prevention After Radiochemotherapy Treatment for Head and Neck Cancer
Acronym: IMPATOX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Collaborators: GORTEC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IMPATOX; VA2009/13 (Other: CRLC Val d'Aurelle-Paul Lamarque)
Record Dates: First submitted 2010-06-22; First posted 2010-06-23 (Estimated); Last update posted 2020-08-13 (Actual); Status verified 2018-12

CONDITIONS: Severe Acute Mucositis; Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Oral immunomodulatory solution (Experimental): The oral supplement is a 74g sachet containing 302 kcal and 16.7g proteins as well as immunonutrients such as L-Arginine, ARN and omega-3.
  Interventions: Dietary Supplement: Oral Impact
- Placebo (Placebo Comparator): The placebo is an identical formula to the Oral Impact but is not enriched with specific nutrients.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Oral Impact — The patients will benefit in each case from a similar energy supplement (either Oral Impact or placebo) during the 5 days preceding the course of chemotherapy. They will receive the supplement 3 times per day at 10am, 3pm and 5pm outside of their meals. In total, the patients will take the supplements for 15 days (3 courses of 5 days). If the patient has difficulty taking the treatment orally, it can be given via an enteral tube (nasogastric tube or percutaneous gastrostomy). All patients in the protocol will systematically receive a dietetic consultation.
  This consultation by a dietician will detect malnutrition and result in nutritional counsel if necessary (advice re. enrichment of diet, CNO without immunonutrients, artificial nutrition). Follow-up appointments with a dietician will be organised every 3 weeks to maintain adherence to the suggested dietary changes.
  Arms: Oral immunomodulatory solution
Dietary Supplement: Placebo — The placebo is an identical formula to the Oral Impact but is not enriched with specific nutrients.
  Arms: Placebo

SUMMARY:
This randomised, double-blind study will compare an oral immunomodulatory solution to a placebo for the prevention of acute severe mucositis in head and neck cancer patients treated surgically and concomitantly with radiochemotherapy. The investigators expect a decrease of 25% of severe acute mucositis in experimental arm.

ELIGIBILITY:
Inclusion Criteria:

* Epidermal carcinoma proven histologically of the sphere ORL (all locations except nasopharynx).
* Patients with tumours of the oral cavity, the oropharynx, the hypopharynx and the larynx treated initially by surgery and eligible for post-operative radio- chemotherapy concomitantly.

NB. The patients with tumours of the larynx or hypopharynx are eligible if the radiotherapy to the oropharyngeal mucosa will be at least 54 Gy and the mucositis can be visualised without the use of instruments.

* Radio-chemotherapy to be given postoperatively.
* Maximum delay of 8 weeks between the operative date and the planned starting date of radio-chemotherapy.
* Performance status (grade OMS): 0, 1, 2
* Nutritional Risk Index ≥ 83.5
* No mucositis.
* Age: 18-75 years
* Life expectancy ≥ 3 months.
* Informed consent obtained from the patient.
* Affiliation with a social security system.

Exclusion Criteria:

* Tumour of nasopharynx
* Mucositis
* Severe sepsis
* Treatment by immunomodulators in the month preceding inclusion
* ATCD allergy to the components of Oral Impact.
* Parenteral nutrition at inclusion
* Usual contraindications to concomitant radio-chemotherapy
* Patient already included in another therapeutic trial involving an experimental molecule
* Female pregnant or susceptible to being pregnant, or breast-feeding. Patient not using appropriate contraceptive measures during the treatment
* Persons deprived of liberty or under guardianship
* Patients unable to commit to the trial schedule for geographical, social or psychological reasons.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2009-11; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
The rate of grade 3 and 4 acute mucosal toxicity | 3 months

SECONDARY OUTCOMES:
Tolerance | through study completion, an average of 3 years
  tolerance of treatment with the CTCAE (Common Terminology Criteria for Adverse Events)
compliance to the oral immunomodulating formula | through study completion, an average of 3 years
overall quality of life (EORTC QLQ-C30 Questionnaire) | through study completion, an average of 3 years
progression-free survival rates | 1, 2 and 3 years
overall survival rates | 1, 2 and 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Institut du Cancer de Montpellier - Val d'Aurelle, Montpellier, France

REFERENCES:
- [Derived] Boisselier P, Kaminsky MC, Thezenas S, Gallocher O, Lavau-Denes S, Garcia-Ramirez M, Alfonsi M, Cupissol D, de Forges H, Janiszewski C, Geoffrois L, Sire C, Senesse P; Head and Neck Oncology and Radiotherapy Group (GORTEC). A double-blind phase III trial of immunomodulating nutritional formula during adjuvant chemoradiotherapy in head and neck cancer patients: IMPATOX. Am J Clin Nutr. 2020 Dec 10;112(6):1523-1531. doi: 10.1093/ajcn/nqaa227. PMID 32936874